CLINICAL TRIAL: NCT00284869
Title: Ethnic Differences in the Inflammatory Response in Systemic Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: EK255/2005
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Endotoxemia
Keywords: LPS; ethnicity; neutrophils; TNF
MeSH Terms: conditions — Endotoxemia

INTERVENTIONS:
Drug: LPS

SUMMARY:
The purpose of this study is to investigate putative ethnic differences in the proinflammatory response in human endotoxemia.

DETAILED DESCRIPTION:
Recent data show that there are significant disparities among genders and races in the incidence of sepsis. While men are consistently more likely to have sepsis than women, the apparent racial disparities are even more striking, approaching a doubling of the risk for sepsis among Afro-Americans. Most prominent is the risk among black men, the group in which sepsis occurs at the youngest age and results in the most deaths. Potential mechanisms for heterogeneous susceptibility to sepsis include genetic differences, which have been explored according to sex but not according to race, and other social and clinical factors.

The goal of this study is to explore whether proinflammatory and procoagulant responses in a well standardised inflammation model are comparable in healthy Caucasian and African volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any trial-related activities. (Trial activities are any procedure that would not have been performed during normal management of the subject).
* Men aged >18 and <40 years
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Treatment with an investigational drug within three weeks prior to this trial
* Participation in an LPS trial within the last 6 weeks
* Hereditary deficiency of protein C or S, or a mutation of FV (Leiden), or any other known abnormality affecting coagulation, fibrinolysis or platelet function
* History of cardiovascular disease
* Liver or kidney dysfunction
* Regular use of medication or alcohol abuse
* Use of any medication within three weeks prior to the first trial day
* Symptoms of a clinically relevant illness in the 3 weeks before the first trial day
* Excessive sporting activities
* Weight over 95 kg

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32
Dates: Start 2006-01; Study Completion 2006-04

PRIMARY OUTCOMES:
neutrophil counts
IL-8
G-CSF

SECONDARY OUTCOMES:
various inflammation and coagulation parameters
Platelets
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christa Firbas, MD, Principal Investigator — Medical University of Vienna, Department of Clinical Pharmacology
Locations (1):
- Medical University of Vienna, Dept. of Clinical Pharmacology, Vienna, Vienna, Austria

REFERENCES:
- [Background] Leitner JM, Firbas C, Mayr FB, Reiter RA, Steinlechner B, Jilma B. Recombinant human antithrombin inhibits thrombin formation and interleukin 6 release in human endotoxemia. Clin Pharmacol Ther. 2006 Jan;79(1):23-34. doi: 10.1016/j.clpt.2005.10.003. PMID 16413239